CLINICAL TRIAL: NCT05128617
Title: Acute Effects of Chemotherapy Administration on Skeletal Muscle of Breast Cancer Patients: the PROTECT-06 Study
Acronym: PROTECT-06
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: Université de Strasbourg - Unité de Recherche 3072 - Mitochondries, Stress oxydant, Protection musculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-004
Record Dates: First submitted 2021-10-04; First posted 2021-11-22 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Protein turnover; Skeletal muscle deconditoning; Breast cancer; Chemotherapy; Muscle biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — EC regimen; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — muscle micro-biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epirubicin-cyclophosphamide: Woman with early breast cancer receiving a first cycle of epirubicin-cyclphosphamide
  Interventions: Drug: Epirubicin-cyclophosphamide
- Paclitaxel: Woman with early breast cancer receiving a first cycle of paclitaxel
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Epirubicin-cyclophosphamide — 1 cycle of Epirubicin-cyclophosphamide
  Other Names: Epirubicin-endoxan
  Groups: Epirubicin-cyclophosphamide
Drug: Paclitaxel — 1 cycle of Paclitaxel
  Other Names: Taxol
  Groups: Paclitaxel

SUMMARY:
Chemotherapy treatments such as epirubicin-cyclophosphamid or paclitaxel lead to severe off-target side effects such as skeletal muscle deconditioning. To date, three different studies investigated skeletal muscle decontioning in breast cancer patients, through long term protocols including all chemotherapy cycle treatment, and highlighted both structural alterations and impaired cellular processes. However, no study is currently availbale on the acute effect of one single chemotherapy administration in breast cancer patients skeletal muscle tissue. Our study is therefore dedicated to the investigation of the acute effect of the first dose administration of both Epuribicin/cyclophosphamide and Paclitaxel chemotherapies on skeletal muscle of breast cancer patients.

DETAILED DESCRIPTION:
Chemotherapy treatments such as epirubicin-cyclophosphamid or paclitaxel lead to severe off-target side effects such as skeletal muscle deconditioning. Resulting from a global perturbation of the muscle homeostasis, skeletal muscle is characterized by both structural and functional alterations that will translate into a decrease in muscle mass and/or force as well as an increase in muscle fatigability. These maladaptations result in a reduced quality of life and an increased treatment-related toxicity, ultimately leading to an increased mortality risk.To date, three different studies investigated skeletal muscle decontioning in breast cancer patients, through long term protocols including all chemotherapy cycle treatment, and highlighted both structural alterations and impaired cellular processes. However, no study is currently availbale on the acute effect of one single chemotherapy administration in breast cancer patients skeletal muscle tissue.Our study is therefore dedicated to the investigation of the acute effect of the first dose administration of both Epuribicin/cyclophosphamide and Paclitaxel chemotherapies on skeletal muscle of breast cancer patients. Our study will particularly explore cellular mechanisms of muscle decontioning, such as protein turnover, mitochondrial homeostasis and fatty infiltrations.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (stade I to III)
* Patient recieving the first administration of epirubicin-cyclophosphamide (group 1) or paclitaxel (group 2) for early breast cancer treatment

Exclusion Criteria:

* History of cancer
* Known chronic pathology
* Pacemaker
* Contraindication to the evaluation of the physical condition
* Contraindication to the local anesthesia for the muscle micro-biopsy
* Breastfeeding or pregnant woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman recieving the first administration of epirubicin-cyclophosphamide (group 1) or paclitaxel (group 2) for early breast cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Investigate the acute effect of chemotherapy administration on protein turnover cellular processes through vastus lateralis biopsies of breast cancer patients | Before and 4 days after the chemotherapy
  Change From Baseline in Western Blots measurements of protein expression levels

SECONDARY OUTCOMES:
Investigate the acute effect of chemotherapy administration on structural alterations | Before and 4 days after the chemotherapy
  Change From Baseline in Cross-Sectional Area (CSA) measurements
Investigate the acute effect of chemotherapy administration on inflammation | Before and 4 days after the chemotherapy
  Change From Baseline in Western Blots measurments of protein expression levels
Investigate the acute effect of chemotherapy administration on mitochondrial homeostasis | Before and 4 days after the chemotherapy
  Change From Baseline in Western Blot measurement of protein expression levels
Investigate the acute effect of chemotherapy administration on fatty infiltrations | Before and 4 days after the chemotherapy
  Change From Baseline in Western Blot measurement of protein expression levels
Investigate the acute effect of chemotherapy administration on satellite cells | Before and 4 days after the chemotherapy
  Change From Baseline in Western Blot measurement of protein expression levels
.Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the skeletal muscle mass | Before and 4 days after the chemotherapy
  Change From Baseline in quantity of muscle mass measured by bioelectrical impedance analysis
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the muscle force | Before and 4 days after the chemotherapy
  Change From Baseline in the maximal isometric strength of the knee with force transducer
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the muscle thickness | Before and 4 days after the chemotherapy
  Change From Baseline in ultrasonography measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the muscle fibers angle of pennation | Before and 4 days after the chemotherapy
  Change From Baseline in ultrasonography measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the muscle fibers fascicle length | Before and 4 days after the chemotherapy
  Change From Baseline in ultrasonography measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the echogenecity | Before and 4 days after the chemotherapy
  Change From Baseline in ultrasonography measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the quality of life | Before and 4 days after the chemotherapy
  Change From Baseline in FACT-G auto-questionnaire measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the appetite loss | Before and 4 days after the chemotherapy
  Change From Baseline in FAACT auto-questionnaire measurement
Comparison of the acute effect of Epirubicin-Cyclophosphamide versus Paclitaxel on the physical activity level | Before and 4 days after the chemotherapy
  Change From Baseline in GPAQ auto-questionnaire measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie Strasbourg Europe, Strasbourg, France